CLINICAL TRIAL: NCT02601105
Title: Topical Centella Asiatica and the Cosmetic Appearance of Stretch Marks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 637397
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Stretch Marks; Striae Distensae; Cosmetic Appearance of Stretch Marks
Keywords: gotu kola; centella asiatica
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Intervention Model Description: 15 patients were enrolled. All 15 patients had one side of abdomen randomized to placebo and one randomized to Centella Asiatica.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Vehicle Cream (Placebo Comparator): Lipoderm® base served as the placebo vehicle control to be applied every night to demarcated 10 x 10 cm area containing stretch marks on randomly assigned side of abdomen for 12 weeks.
  Interventions: Other: Placebo Vehicle Cream
- Centella Asiatica Cream (Experimental): An alcoholic extract of CA (verified by HPLC) mixed into a Lipoderm® base served as the treatment cream to be applied every night to demarcated 10 x 10 cm area containing stretch marks on the opposite side of the abdomen for 12 weeks.
  Interventions: Other: Centella Asiatica Cream

INTERVENTIONS:
Other: Placebo Vehicle Cream — Lipoderm Cream alone
  Arms: Placebo Vehicle Cream
Other: Centella Asiatica Cream — 1% Centella Asiatica in lipoderm
  Arms: Centella Asiatica Cream

SUMMARY:
The purpose of this study is to clinically evaluate the efficacy, safety as well as patient satisfaction in the use of topical Centella asiatica (CA) on the cosmetic appearance of stretch marks.

DETAILED DESCRIPTION:
Subjects with abdominal stretch marks will be enrolled in to this study. The presence of abdominal stretch marks will be confirmed by a board certified dermatologist. The right and the left side of the abdomen will be randomized by binary randomization to treatment with CA cream or the vehicle cream. Therefore each patient will serve as their own control.

Each half of the abdomen will be subjected to topical treatment with CA 1% Cream formulated in PCCA Lipoderm® base or PCCA Lipoderm® base as the placebo vehicle treatment based on prior randomization. The creams will be given to the patient in blinded fashion: Cream A (containing CA) and cream B (vehicle/placebo) with instructions apply both formulations daily at night.

Patients will be asked to return to clinic at 6 weeks and 12 weeks for follow up assessment for a total of 3 sessions (baseline, 6 weeks, 12 weeks). High-resolution digital photographs of the stretch marks will be taken at baseline and at each follow-up visit to document clinical response. Two physician graders blinded to the photographs and the treatments will assess cosmetic outcome on a six-point analog scale

The width of the treated stretch marks in each subject will also be measured at the baseline and 8 weeks after the final treatment. The difference of the width will be converted into the percentage of reduction from the baseline.

Subjects will also be asked to complete two surveys at each visit. The two surveys include patient satisfaction with cosmetic and clinical outcome based on a five-point scale.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking subjects over the age of 18
2. Subjects clinically diagnosed with stretch marks

Exclusion Criteria:

1. History of keloid scarring
2. Isotretinoin use within the last 6 months
3. Oral prednisone use within the last 3 months
4. Non-ablative laser procedures to the abdomen within 1 year of study initiation
5. Ablative resurfacing procedures to the abdomen within 3 years of the study initiation
6. Pregnancy
7. Use of immunosuppressive drugs
8. Known hypersensitivity to Centella asiatica

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, MS, CAT, Principal Investigator — UC Davis Department of Dermatology
Locations (1):
- University of California Davis, Sacramento, California, United States

REFERENCES:
- [Background] Cho S, Park ES, Lee DH, Li K, Chung JH. Clinical features and risk factors for striae distensae in Korean adolescents. J Eur Acad Dermatol Venereol. 2006 Oct;20(9):1108-13. doi: 10.1111/j.1468-3083.2006.01747.x. PMID 16987267
- [Background] Brinkhaus B, Lindner M, Schuppan D, Hahn EG. Chemical, pharmacological and clinical profile of the East Asian medical plant Centella asiatica. Phytomedicine. 2000 Oct;7(5):427-48. doi: 10.1016/s0944-7113(00)80065-3. PMID 11081995
- [Background] Incandela L, Cesarone MR, Cacchio M, De Sanctis MT, Santavenere C, D'Auro MG, Bucci M, Belcaro G. Total triterpenic fraction of Centella asiatica in chronic venous insufficiency and in high-perfusion microangiopathy. Angiology. 2001 Oct;52 Suppl 2:S9-13. PMID 11666128
- [Background] Lu L, Ying K, Wei S, Fang Y, Liu Y, Lin H, Ma L, Mao Y. Asiaticoside induction for cell-cycle progression, proliferation and collagen synthesis in human dermal fibroblasts. Int J Dermatol. 2004 Nov;43(11):801-7. doi: 10.1111/j.1365-4632.2004.02047.x. PMID 15533060
- [Background] Rosen H, Blumenthal A, McCallum J. Effect of asiaticoside on wound healing in the rat. Proc Soc Exp Biol Med. 1967 May;125(1):279-80. doi: 10.3181/00379727-125-32070. No abstract available. PMID 6027541
- [Background] Sunilkumar, Parameshwaraiah S, Shivakumar HG. Evaluation of topical formulations of aqueous extract of Centella asiatica on open wounds in rats. Indian J Exp Biol. 1998 Jun;36(6):569-72. PMID 9731470
- [Result] Gungor S, Sayilgan T, Gokdemir G, Ozcan D. Evaluation of an ablative and non-ablative laser procedure in the treatment of striae distensae. Indian J Dermatol Venereol Leprol. 2014 Sep-Oct;80(5):409-12. doi: 10.4103/0378-6323.140296. PMID 25201840
- [Result] Mazzarello V, Farace F, Ena P, Fenu G, Mulas P, Piu L, Rubino C. A superficial texture analysis of 70% glycolic acid topical therapy and striae distensae. Plast Reconstr Surg. 2012 Mar;129(3):589e-590e. doi: 10.1097/PRS.0b013e3182419c40. No abstract available. PMID 22374035
- [Result] Garcia Hernandez JA, Madera Gonzalez D, Padilla Castillo M, Figueras Falcon T. Use of a specific anti-stretch mark cream for preventing or reducing the severity of striae gravidarum. Randomized, double-blind, controlled trial. Int J Cosmet Sci. 2013 Jun;35(3):233-7. doi: 10.1111/ics.12029. Epub 2013 Jan 15. PMID 23237514

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The right and the left side of the abdomen were randomized by binary randomization to treatment with CA cream or the vehicle cream. Therefore each patient will serve as their own control.
Groups:
- All Study Participants: Placebo Vehicle Cream: Lipoderm Cream Alone Lipoderm® base served as the placebo vehicle control to be applied every night to demarcated 10 x 10 cm area containing stretch marks on randomly assigned side of abdomen for 12 weeks.
  Centella Asiatica: 1% Centella Asiatica in Lipoderm Cream An alcoholic extract of CA (verified by HPLC) mixed into a Lipoderm® base served as the treatment cream to be applied every night to demarcated 10 x 10 cm area containing stretch marks on the opposite side of the abdomen for 12 weeks.
Period: Placebo Cream; Centella Asiatica Bsln.
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Placebo Cream; Centella Asiatica Week 6
Arm/Group | All Study Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Placebo Cream; Centella Asiatica Week 12
Arm/Group | All Study Participants
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The right and the left side of the abdomen were randomized by binary randomization to treatment with CA cream or the vehicle cream. Therefore each patient will serve as their own control.
Units Other Than Participants: Side of Abdomen
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Number analyzed (Side of Abdomen) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.5 [24 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Cosmetic Outcome- Fraction Improving by at Least 1 Point Increase in Overall Appearance of Stretch Marks
Description: Assessed by four blinded evaluators by observing comparative baseline photographs using 6 point scale (worsened = -1 points, no improvement = 0 points, mild = 1 points, <25% improvement, moderate = 2 points, 26-50% improvement, good = 3 points, 51-75% improvement, excellent = 4 points, >75% improvement)
Time Frame: 12 weeks
Population: 13 participants completed all study procedures and were included in data analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Vehicle Cream: Lipoderm® base served as the placebo vehicle control to be applied every night to demarcated 10 x 10 cm area containing stretch marks on randomly assigned side of abdomen for 12 weeks.
  Placebo Vehicle Cream: Lipoderm cream
- Centella Asiatica: An alcoholic extract of CA (verified by HPLC) mixed into a Lipoderm® base served as the treatment cream to be applied every night to demarcated 10 x 10 cm area containing stretch marks on the opposite side of the abdomen for 12 weeks.
  Centella Asiatica: 1% Centella Asiatica in lipoderm
Arm/Group | Placebo Vehicle Cream | Centella Asiatica
Number analyzed (Participants) | 13 | 13
Participants | 3 | 5

2. Primary Outcome: Stretch Mark Width/Area
Description: Stretch mark width: measured at week 12. This will be converted into the percentage of reduction from the baseline.
Time Frame: 12 weeks
Population: 13 participants completed all study procedures and were included in data analysis.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Vehicle Cream | Centella Asiatica
Number analyzed (Participants) | 13 | 13
percent change | 0.8 (0.05) | 0.87 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the study duration of 12 weeks.
Arm/Group | Placebo Vehicle Cream | Centella Asiatica
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No